CLINICAL TRIAL: NCT04609982
Title: Randomized Controlled Trial Evaluating the Impact of Noise Exposure in Otolaryngology Floor Among Head and Neck Cancer Patients
Brief Title: SSNHL in Head & Neck Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI did not respond to the REBs concerns and they closed the study
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1025581
Record Dates: First submitted 2020-10-15; First posted 2020-10-30 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Ear Protective Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wearing ear plugs (Experimental)
  Interventions: Device: ear plugs
- Not wearing ear drops (No Intervention)

INTERVENTIONS:
Device: ear plugs — giving half of the patients ear plugs
  Arms: wearing ear plugs

SUMMARY:
A sound dosimeter will be used to measure noise level to which a population of head and neck patients on the otolaryngology ward are exposed to. The device is the EXTECH 407764 type II sound level meter (IEC 651 RS232). The device will be configured to OSHA and ISO standards, and calibration confirmed in a sound booth with a sound level calibrator. The dosimeter captures A-weighted sound levels between 30 and 130 dB. Specifically, participants included in the study will be head and neck cancer patients on the otolaryngology floor at VG site. Measurements will be taken three times a day at random intervals. Each measurement will be taken in a similar manner. The dosimeter will be placed on the head side of the bed at the level of patient's ear one inch away from the ear and kept there for ten seconds to get a representative level. The overall measurements will be averaged (Leq) for statistical analysis. Investigators will randomly select 50% of the patients and give them protective ear plugs to be used while the participants are inpatients, and the other 50% will not provide them with ear plugs (like what is being done now). Investigators will obtain a baseline hearing test prior to admission and 7 days after admission and then a repeat hearing test at 3 weeks after discharge. The goal is to establish if there is a temporary or a permanent threshold shift.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnoses of head and neck disease requiring surgery.
* Must be expected to be admitted to ENT floor.
* Must be able to conduct a hearing test.

Exclusion Criteria:

* a diagnoses of SNHL.
* participants with low mental capacity.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-20 (Estimated); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-11-20 (Estimated)

PRIMARY OUTCOMES:
Hearing loss | 6 months
  investigators will measure the level hearing loss during the patients stay using a hearing test done by an audiologist. the rate level of hearing loss will be measured by dB using an audiogram.

IPD SHARING:
Plan to Share IPD: No